CLINICAL TRIAL: NCT03944603
Title: Investigating the Contribution of Peripheral Versus Central Nervous System Dysfunction to Cognitive Aging
Brief Title: Longitudinal Innate Immunity and Aging Study
Acronym: LIIA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-2607; R01AG058772 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-05-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy Older Adults Ages 60-89
Keywords: Alzheimer's Disease; Dementia; Older Adult; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Alzheimer Disease; Dementia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study plans to examine biological bases of cognitive aging. The goals of the study are to better understand how immune system markers, measured in the blood and in the spinal fluid, are related to clinical features of aging over time. The study also aims to better understand how different types of biomarkers may relate to immune health and the aging process. This research may ultimately help us better understand what puts individuals at risk for cognitive decline and for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages of 60-89
2. Have a reliable study partner who has frequent contact with the subject (i.e., at least twice per month) and is able to provide information about functional abilities
3. Mini Mental State Examination (MMSE) >23
4. Clinical Dementia Rating (CDR) global score of 0
5. No informant report of significant cognitive decline in prior year
6. No evidence from the screening visit suggesting a neurodegenerative disorder (per team neurologist)
7. Willingness to complete both baseline and 2-year follow-up procedures

Exclusion Criteria:

1. Major psychiatric disorder (e.g. schizophrenia, bipolar disorder, untreated major depression within past year)
2. Neurological conditions affecting cognition (e.g. Parkinson's disease, epilepsy (onset prior than 2 years ago), head trauma with loss of consciousness >5 min within past two years, large vessel infarct, mild cognitive impairment, or dementia)
3. CNS immune conditions and other conditions affecting cognition (e.g., multiple sclerosis, paraneoplastic encephalitides; Hashimoto's encephalopathy; systematic lupus erythematosus)
4. Systematic illness (e.g.,current cancer, renal failure, respiratory failure)
5. Substance abuse/dependence (DSM-V criteria)
6. Current medication use likely to affect CNS (e.g., long-acting benzodiazepines, neuroleptics in the phenothiazine and haloperidol families)
7. Current medication use that precludes lumbar punctures (e.g. anticoagulants, antiplatelets, heparin shots, or some other blood thinner medications: Warfarin [coumadin], Pradaxa [dabigatran], Xarelto [rivaroxaban]. Eliquis [apixaban], or Plavix [clopidogrel].
8. Significant sensory or motor deficits that would interfere with cognitive testing
9. Factors that preclude MR imaging (e.g., pacemaker)
10. Factors that preclude lumbar puncture

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Levels of Immune Protein Markers in Blood and CSF | 2-Year Changes
  Outcome measures will include longitudinal changes in protein levels of blood inflammation and CSF inflammation
Performance on Neuropsychological Measures | 2-Year Changes
  Outcome measures will include longitudinal changes in cognitive measures (e.g., memory and executive functions) over time
Levels of Exosomal Innate Immune Markers in Blood and CSF | 2-Year Changes
  Outcome measures will include longitudinal changes in innate immune markers in exosomes (i.e., extracellular vesicles)

SECONDARY OUTCOMES:
Brain Structure | Baseline
  Outcome measures will include baseline structural brain imaging
CSF Levels of Alzheimer's Disease Related Markers | 2-year change
  Outcome measures will include CSF levels of proteins associated with Alzheimer's disease pathology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No